CLINICAL TRIAL: NCT04574570
Title: Clinical Evaluations of the TOKA Customized Device for High Tibial Osteotomy in the Treatment of Knee Osteoarthritis: a Pilot Study.
Brief Title: TOKA: Custom Made Devices for High Tibial Osteotomy (HTO) - Clinical Investigation
Acronym: TOKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3D Metal Printing Ltd (Industry)
Collaborators: University of Bath (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE-AVEC 623/2019 DISP/IOR TOKA
Record Dates: First submitted 2020-09-10; First posted 2020-10-05 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2024-02

CONDITIONS: Unicompartmental Medial Knee Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional patient (Other): Personalised High Tibial Osteotomy (HTO) using a patient-specific fixation plate (TOKA®)
  Interventions: Device: High Tibial Osteotomy

INTERVENTIONS:
Device: High Tibial Osteotomy — Personalised High Tibial Osteotomy (HTO) using a patient-specific fixation plate (TOKA®)

SUMMARY:
This preliminary pilot study is a single-centre, prospective, uncontrolled, 32-month study to assess the performance of personalised opening wedge High Tibial Osteotomy (HTO) treatment using the TOKA® device and procedure.

The medical device being examined is a custom-made device and therefore does not require a CE mark. Furthermore, the study will serve as a useful method of gathering clinical data and measuring device performance, as well as establishing a potential commercial relationship with the hospital administration.

Study Objectives::

1. to assess the morphology of the knee joint and the improvement of OA following the TOKA® treatment.
2. to Assess the functional outcome of the knee joint and the improvement of OA following the TOKA® treatment.

Outcomes Evaluations::

1. The morphology of the knee joint is assessed by verifying the matching between the planned correction and the post-operative imaging results, along with the investigation of the maintenance of the desired correction at the follow-up meetings. These results are measured through the correction angle, hip-knee-ankle angle (HKA - mechanical axis), Mikulicz point (recorded as a percentage of the tibial width from the medial to the lateral region) and posterior slope, using the imaging techniques.
2. The functional outcome of the knee joint is assessed by a) performing a gait analysis of the patients pre-operatively and post-operatively, b) the use of clinical scoring...

   .

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing opening wedge Hight Tibial Osteotomy (HTO)
* Patients must have completed a consent form for the study
* Patients must be prepared to comply with the pre and post-operative investigations, rehabilitation, attendance schedule and questionnaire schedule of the study
* Patient in whom any varus deformity present is <20°
* The diagnosis is of unicompartmental medial osteoarthritis of the knee
* Patient has primary diagnosis of Non-Inflammatory Degenerative Joint Disease (NIDJD)
* BMI<40
* Age range 40 to 65 years

Exclusion Criteria:

* Refusal to consent to the study
* Pregnancy
* Prisoners
* A patient known to have substance abuse or psychological disorders that could interfere with their ability to comply with the post-operative rehabilitation and assessment schedules
* Patients unable to read or understand the patient information leaflet and consent form
* Patient has a known sensitivity to device materials.
* Patient has a Body Mass Index (BMI) ≥ 40.
* Patient has an active or suspected latent infection in or about the affected knee joint at time of study device implantation.
* Patient has received any orthopaedic surgical intervention to the lower extremities within the past year or is expected to require any orthopaedic surgical intervention to the lower extremities, other than the HTO to be enrolled in this study, within the next year.
* Patient requires bilateral HTO or has a history of unsuccessful contralateral partial replacement or HTO.
* Patient has chronic heart failure (NYHA Stage ≥ 2)
* Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device.
* Patient is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's disease) leading to progressive bone deterioration.
* Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akizuki S, Shibakawa A, Takizawa T, Yamazaki I, Horiuchi H. The long-term outcome of high tibial osteotomy: a ten- to 20-year follow-up. J Bone Joint Surg Br. 2008 May;90(5):592-6. doi: 10.1302/0301-620X.90B5.20386. PMID 18450624
- [Background] Bedson J, Croft PR. The discordance between clinical and radiographic knee osteoarthritis: a systematic search and summary of the literature. BMC Musculoskelet Disord. 2008 Sep 2;9:116. doi: 10.1186/1471-2474-9-116. PMID 18764949
- [Background] Elson DW, Petheram TG, Dawson MJ. High reliability in digital planning of medial opening wedge high tibial osteotomy, using Miniaci's method. Knee Surg Sports Traumatol Arthrosc. 2015 Jul;23(7):2041-8. doi: 10.1007/s00167-014-2920-x. Epub 2014 Mar 1. PMID 24584646
- [Background] Ren YM, Duan YH, Sun YB, Yang T, Hou WY, Zhu RS, Tian MQ. Opening-Wedge High Tibial Osteotomy Using Autograft versus Allograft: A Systematic Review and Meta-analysis. J Knee Surg. 2020 Jun;33(6):565-575. doi: 10.1055/s-0039-1681065. Epub 2019 Mar 12. PMID 30861539
- [Background] Harris JD, McNeilan R, Siston RA, Flanigan DC. Survival and clinical outcome of isolated high tibial osteotomy and combined biological knee reconstruction. Knee. 2013 Jun;20(3):154-61. doi: 10.1016/j.knee.2012.12.012. Epub 2013 Mar 9. PMID 23477914
- [Background] Kallala RF, Vanhegan IS, Ibrahim MS, Sarmah S, Haddad FS. Financial analysis of revision knee surgery based on NHS tariffs and hospital costs: does it pay to provide a revision service? Bone Joint J. 2015 Feb;97-B(2):197-201. doi: 10.1302/0301-620X.97B2.33707. PMID 25628282
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Konopka JF, Gomoll AH, Thornhill TS, Katz JN, Losina E. The cost-effectiveness of surgical treatment of medial unicompartmental knee osteoarthritis in younger patients: a computer model-based evaluation. J Bone Joint Surg Am. 2015 May 20;97(10):807-17. doi: 10.2106/JBJS.N.00925. PMID 25995491
- [Background] Niinimaki TT, Eskelinen A, Mann BS, Junnila M, Ohtonen P, Leppilahti J. Survivorship of high tibial osteotomy in the treatment of osteoarthritis of the knee: Finnish registry-based study of 3195 knees. J Bone Joint Surg Br. 2012 Nov;94(11):1517-21. doi: 10.1302/0301-620X.94B11.29601. PMID 23109632
- [Background] Smith WB 2nd, Steinberg J, Scholtes S, Mcnamara IR. Medial compartment knee osteoarthritis: age-stratified cost-effectiveness of total knee arthroplasty, unicompartmental knee arthroplasty, and high tibial osteotomy. Knee Surg Sports Traumatol Arthrosc. 2017 Mar;25(3):924-933. doi: 10.1007/s00167-015-3821-3. Epub 2015 Oct 31. PMID 26520646
- [Background] Verra WC, Witteveen KQ, Maier AB, Gademan MG, van der Linden HM, Nelissen RG. The reason why orthopaedic surgeons perform total knee replacement: results of a randomised study using case vignettes. Knee Surg Sports Traumatol Arthrosc. 2016 Aug;24(8):2697-703. doi: 10.1007/s00167-015-3961-5. Epub 2016 Jan 12. PMID 26759152
- [Derived] Zaffagnini S, Dal Fabbro G, Lucidi GA, Agostinone P, Belvedere C, Leardini A, Grassi A. Personalised opening wedge high tibial osteotomy with patient-specific plates and instrumentation accurately controls coronal correction and posterior slope: Results from a prospective first case series. Knee. 2023 Oct;44:89-99. doi: 10.1016/j.knee.2023.07.011. Epub 2023 Aug 8. PMID 37562120
- [Derived] Ruggeri M, Gill HS, Leardini A, Zaffagnini S, MacLeod A, Ortolani M, Faccia F, Grassi A, Fabbro GD, Durante S, Belvedere C. Superimposition of ground reaction force on tibial-plateau supporting diagnostics and post-operative evaluations in high-tibial osteotomy. A novel methodology. Gait Posture. 2022 May;94:144-152. doi: 10.1016/j.gaitpost.2022.02.028. Epub 2022 Feb 25. PMID 35334334

RESULTS

PARTICIPANT FLOW:
Groups:
- Interventional Patient: Patients selected and operated for personalised High Tibial Ostotomy (HTO) using theTOKA®
Period: Overall Study
Arm/Group | Interventional Patient
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 25
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 26.8 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Morphology Assessment Via Correction Angle Assessment
Description: The device morphology assessment is performed by verifying the matching between the planned correction and the post-operative imaging results, along with the investigation of the maintenance of the desired correction at the follow-up meetings. These results are measured through the correction angle, using image-based techniques.
Time Frame: At 6 months after surgery
Population: Operated Patients
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
Degree | 1.5 (2.0)

2. Primary Outcome: Morphology Assessment Via Hip-knee-ankle Angle Assessment
Description: The device morphology assessment is performed by verifying the matching between the planned correction and the post-operative imaging results, along with the investigation of the maintenance of the desired correction at the follow-up meetings. These results are measured through the hip-knee-ankle angle (HKA - mechanical axis) reported in degree, using image-based techniques.
Time Frame: At 6 months after surgery
Population: Operated patients
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
Degree | 1.5 (2.0)

3. Primary Outcome: Morphology Assessment Via Mikulicz Point Assessment
Description: The device morphology assessment is performed by verifying the matching between the planned correction and the post-operative imaging results, along with the investigation of the maintenance of the desired correction at the follow-up meetings. These results are measured through the Mikulicz point reported in % of the tibial width from the medial to the lateral region, using image-based techniques.
Time Frame: At 6 months after surgery
Measure: Mean (Standard Deviation); unit: % of medial-lateral tibial plateau width
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
% of medial-lateral tibial plateau width | -9.7 (8.4)

4. Primary Outcome: Morphology Assessment Via Posterior Slope Assessment
Description: The device morphology assessment is performed by verifying the matching between the planned correction and the post-operative imaging results, along with the investigation of the maintenance of the desired correction at the follow-up meetings. These results are measured through the posterior slope reported in degree, using image-based techniques.
Time Frame: At 6 months after surgery
Population: Operated patiemts
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
Degree | 0.1 (0.3)

5. Secondary Outcome: Functional Assessment Via Gait Analysis - Kinematics
Description: The functional assessment is performed via three dimensional gait analysis of the patients before surgery. Relevant kinematic results are reported in terms of joint rotations (in degrees)..
Time Frame: Before surgery
Population: Operated Patients - Max Knee Flexion Rotation
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
Degree | 70.5 (5.0)

6. Secondary Outcome: Functional Assessment Via Gait Analysis - Kinetics
Description: The functional assessment is performed via three dimensional gait analysis of the patients before surgery. Relevant kinetic results are reported in terms of joint moments (in N*mm, normalized to patient's body weight times height).
Time Frame: Before surgery
Population: Operated Patients - Max Abduction Moment
Measure: Mean (Standard Deviation); unit: % of Body Weight * height
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
% of Body Weight * height | 3.8 (1.2)

7. Secondary Outcome: Functional Assessment Via Clinical Scoring - Knee Osteoarthritis Outcome Score
Description: The functional assessment is performed via clinical scoring using the Knee Osteoarthritis Outcome Score (KOOS). KOOS value range: [min / max]= 0 - 100, higher values mean better outcome.
Time Frame: 6 months after surgery.
Population: Operated patients - KOOS (total) at 6 month after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
score on a scale | 81.2 (9.7)

8. Secondary Outcome: Functional Assessment Via Clinical Scoring - European Quality of Life Via 5-Dimensions Questionnaire
Description: The functional assessment is performed via clinical scoring using the European Quality of life via 5-Dimensions questionnaire (EQ-5D). In this applied scoring system, respondents rank their health status into 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension can be rated from 1 to 3 as follows: 1=no problem, 2=moderate problems or 3=severe problems.
  The final total score is the sum of the scores given to each dimension and ranges from 5 (best outcome) to 15 (worst outcome).
Time Frame: 6 months after surgery.
Population: Operated patients - European Quality of life via 5-Dimensions questionnaire (total) at 6 month after surgery
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
units on scale | 7.5 (0.9)

9. Secondary Outcome: Functional Assessment Via Clinical Scoring - Tegner Score
Description: The functional assessment is performed via clinical scoring using the Tegner score. Tegner scale value range: [min / max]= 0 - 10, higher values mean better outcome.
Time Frame: 6 month after surgery.
Population: Pot operative patients at 6 month after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
score on a scale | 4.2 (1.3)

10. Secondary Outcome: Functional Assessment Via Clinical Scoring - Knee Society System Score
Description: The functional assessment is performed via clinical scoring using the knee society system score (KSS). KSS value range: [min / max]= 0 - 100, higher values mean better outcome.
Time Frame: 6 months after surgery.
Population: Operated patients - KSS (total) at 6 months after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
score on a scale | 93.5 (13.7)

11. Secondary Outcome: Functional Assessment Via Clinical Scoring - Visual Analogue Scale
Description: The functional assessment is performed via clinical scoring using the Visual Analogue Scale (VAS). VAS is based on a 10-cm long straight line with one end meaning no pain and the other end meaning the worst pain.
  The score is from 0 to 10 (0= no pain, 10= worst pain ever)
Time Frame: 6 months after surgery.
Population: Operated patients - VAS at 6 month after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
score on a scale | 1.3 (1.0)

12. Secondary Outcome: The Functional Assessment Via X-ray Examinations
Description: The functional assessment is performed via x-ray examinations by reporting knee joint alligments in degrees..
Time Frame: Before surgery and at 1, 3, 6, 12 and 24 months after surgery.
Population: Operated patients at 6 months after surgery
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
Degree | 181.9 (2.6)

13. Secondary Outcome: Functional Assessment Via Gait Analysis - Kinematics
Description: The functional assessment is performed via three dimensional gait analysis of the patients before and after surgery. Relevant kinematic results are reported in terms of joint rotations (in degrees)..
Time Frame: 6 months after surgery
Population: Operated Patients - Max Knee Flexion Rotation at 6 months after surgery
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
Degree | 58 (6.0)

14. Secondary Outcome: Functional Assessment Via Gait Analysis - Kinetics
Description: The functional assessment is performed via three dimensional gait analysis of the patients before and after surgery. Relevant kinematic results are reported in terms of joint moments (in N*mm, normalized to patient's body weight times height).
Time Frame: at 6 months after surgery
Population: Operated Patients - Max Abduction Moment
Measure: Mean (Standard Deviation); unit: % of Body Weight * height
Arm/Group | Interventional Patient
Number analyzed (Participants) | 25
% of Body Weight * height | 2.8 (0.8)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Interventional Patient
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT04574570/Prot_002.pdf
  • Informed Consent Form (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT04574570/ICF_000.pdf